CLINICAL TRIAL: NCT05175885
Title: Multicenter, Prospective and Open-label Clinical Trial to Evaluate the Viability, Performance and Safety of ex Vivo Normothermic Perfusion in Kidney Transplantation From DCD and DBD Donors.
Brief Title: Ex Vivo Normothermic Perfusion in Kidney Transplantation.
Acronym: KidneyARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ebers Medical Technology, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KidneyARK
Record Dates: First submitted 2021-12-02; First posted 2022-01-04 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Transplantation; EBERS; EVNP; Ex vivo normothermic perfusion; DCD; DBD; Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function | interventions — Cryopreservation

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective and open-label clinical investigation to evaluate the viability, performance and safety of ex vivo normothermic perfusion in kidney transplantation from DCD and DBD donors and compare it by means of retrospective matching with static cold storage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Ex vivo normothermic perfusion (EVNP) of the graft with the Ark Kidney System
  Interventions: Device: Ex vivo normothermic perfusion
- Historical control group (Active Comparator): Nonrandomized historical control group formed by patients transplanted without ex vivo normothermic perfusion (EVNP) in the period Sept 2015-Sept 2020, selected by retrospective matching.
  Interventions: Device: Cold preservation

INTERVENTIONS:
Device: Ex vivo normothermic perfusion — Ex vivo normothermic perfusion (EVNP) of the renal graft with the Ark Kidney System
  Other Names: EVNP
  Arms: Experimental group
Device: Cold preservation — Static cold storage (SCS) or hypothermic machine perfusion (HMP) of the renal graft
  Other Names: SCS/HMP
  Arms: Historical control group

SUMMARY:
A multicenter, prospective and open-label clinical investigation to evaluate the viability, performance and safety of ex vivo normothermic perfusion in kidney transplantation from DCD and DBD donors.

DETAILED DESCRIPTION:
The Ark Kidney is a medical device for ex vivo normothermic perfusion intended to create the conditions that allow kidneys to be resuscitated and / or preserved prior to transplantation. It consists of a permanent unit, which is retained after each perfusion, and a disposable circuit called the ARK Kidney Kidney Disposable Set (KDS), which must be replaced after perfusion to ensure sterile conditions.

It is a portable organ perfusion system designed to preserve a kidney by continuous perfusion of the donated organ with warm oxygenated perfusate supplemented with erythrocytes from the blood bank. The perfusion solution circulates continuously through the vascular network of the organ in a closed circuit. During perfusion, the system can monitor organ perfusion parameters, as well as the conditions of the perfusion solutions and the volume of urine generated during the perfusion.

The primary objective of the clinical study is to assess the viability, performance and safety of ex vivo normothermic perfusion with the Ark Kidney in kidney transplantation from DCD and DBD donors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and older
2. Patients undergoing renal replacement therapy by means of dialysis and included in the waiting list for renal transplantation in their respective site.
3. Candidates to receive a first or second renal transplant from (i) a Maastricht type III (Maastricht classification) controlled DCD donor or (ii) a DBD donor aged 70 years or older.
4. Patients that have given informed consent in written form before their inclusion in the study. In case of compromised mental capacity, the approval and signature of a legal guardian will be required.
5. Patients compliant with the requirements of the study and without impediments to follow the instructions throughout the 1-year duration of the study.
6. Patients that meet the acceptance criteria for kidney transplant recipients established in the clinical site in agreement with usual clinical practice.

Exclusion Criteria:

1. Two or more previous kidney transplantations
2. Dual kidney transplantation or multivisceral transplantation (e.g. a pancreas-kidney transplantation)
3. Recipients of an organ with any of the following characteristics:

   1. Expected cold ischemia time before EVNP > 20 hours
   2. Organ from hepatitis B surface antigen-positive or hepatitis C viremic donor
   3. Organ with multiple arteries
4. Recipients with body mass index (BMI) > 40 kg/m2
5. Diagnosis of focal segmental glomerulosclerosis (FSGS) or membranoproliferative glomerulonephritis with high recurrence risk after transplantation in the eyes of the investigator.
6. Diagnosis of atypical hemolytic-uremic syndrome or thrombotic microangiopathy at the moment of inclusion
7. Diagnosis of antiphospholipid syndrome at the moment of inclusion
8. Panel-reactive antibodies (PRA) score > 50%
9. Known allergies to any of the components of the perfusate
10. Preexisting vascular disease that represents an extraordinary technical difficulty for the transplantation in the opinion of the investigator
11. Presence of clinically relevant donor-specific anti-HLA antibodies
12. ABO incompatibility
13. History of alcohol or drug abuse in the last two years
14. Use of normothermic regional perfusion during the organ harvesting process
15. Participation of the patient in another study or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety of EVNP in kidney transplantation from DCD and DBD donors as evaluated by assessment of adverse events | 1 year
  The rate of adverse events will be compared in intervention arm and control arm

SECONDARY OUTCOMES:
Delayed graft function (DGF) | 1 week
  Delayed graft function (DGF), defined as the need for dialysis during the first week after transplantation
Duration (in days) of delayed graft function (DGF) | 1 month
  Duration (in days) of delayed graft function (DGF)
Proportion of patients with functional delayed graft function (fDGF) | 1 week
  Proportion of patients with functional delayed graft function (fDGF), defined as the failure of serum creatinine to decrease by at least 10% daily on 3 consecutive days during the first week post-transplant, without need for dialysis in that time.
Primary non-function (PNF) | 1 week
  Primary non-function (PNF)
Graft renal function (1 day) | 1 day
  Graft renal function, measured by the levels of serum creatinine and eGFR (CKD-EPI) at day 1 post-transplant in recipients who have not gone through dialysis after transplantation.
Graft renal function (3 days) | 3 days
  Graft renal function, measured by the levels of serum creatinine and eGFR (CKD-EPI) at day 3 post-transplant in recipients who have not gone through dialysis after transplantation.
Graft renal function (5 days) | 5 days
  Graft renal function, measured by the levels of serum creatinine and eGFR (CKD-EPI) at day 5 post-transplant in recipients who have not gone through dialysis in the previous three days.
Graft renal function (7 days) | 7 days
  Graft renal function, measured by the levels of serum creatinine and eGFR (CKD-EPI) at day 7 post-transplant in recipients who have not gone through dialysis in the previous three days.
Graft renal function (30 days) | 30 days
  Graft renal function, measured by the levels of serum creatinine and eGFR (CKD-EPI) at day 30 post-transplant in recipients who have not gone through dialysis in the previous three days.
Graft renal function (90 days) | 90 days
  Graft renal function, measured by the levels of serum creatinine and eGFR (CKD-EPI) at day 90 post-transplant in recipients who have not gone through dialysis in the previous three days.
Patient survival | 1 year
  Patient survival
Graft survival | 1 year
  Graft survival
Performance of EVNP in kidney transplantation from DCD and DBD donors as evaluated by the fraction of non-implanted organs because of the preservation method | 1 day
  The fraction of non-implanted organs will be compared in intervention arm and control arm
Viability of EVNP in kidney transplantation from DCD and DBD donors as evaluated by the ratio of planned vs. perfused organs | 1 day
  Viability of EVNP will be determined by the ratio of planned vs. perfused organs

CONTACTS AND LOCATIONS:
Overall Officials: Alex Gutierrez-Dalmau, MD, Principal Investigator — Miguel Servet University Hospital
Locations (1):
- Miguel Servet University Hospital, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No